CLINICAL TRIAL: NCT01706315
Title: A Randomized, Single Blind, Placebo-Controlled Study to Evaluate Safety, Tolerability, and Pharmacokinetics of Repeat Escalating Oral Doses of GSK2140944 in Healthy Adult Subjects (BTZ116778)
Brief Title: This Study Will Investigate the Safety, Tolerability and Pharmacokinetic Profile of Repeat Oral Doses of GSK2140944 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 116778
Record Dates: First submitted 2012-10-11; First posted 2012-10-15 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Infections, Respiratory Tract
MeSH Terms: conditions — Respiratory Tract Infections | interventions — gepotidacin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (12):
- Cohort 1 - GSK2140944 400 mg (Experimental): Subjects will be randomized in 6:2 ratio to receive either GSK2140944 (Day 1: Single oral dose Days 3 to 16: (14 Days) BID oral doses) or placebo for approximately 15 days
  Interventions: Drug: GSK2140944
- Cohort 1 - Placebo (Placebo Comparator): Subjects will be randomized in 6:2 ratio to receive either GSK2140944 BID or matching placebo for approximately 15 days
  Interventions: Drug: Placebo
- Cohort 2 - GSK2140944 800 mg (Experimental): Subjects will be randomized in 12:4 ratio to receive either GSK2140944 (Day 1: Single oral dose Days 3 to 16: (14 Days) BID oral doses) or placebo for approximately 15 days. GSK2140944 dose in Cohort 2 will be decided based on the safety and PK data from six subjects in Cohort 1
  Interventions: Drug: GSK2140944
- Cohort 2 - Placebo (Placebo Comparator): Subjects will be randomized in 12:4 ratio to receive either GSK2140944 BID or matching placebo for approximately 15 days
  Interventions: Drug: Placebo
- Cohort 3 - GSK2140944 1500 mg (Experimental): Subjects will be randomized in 12:4 ratio to receive either GSK2140944 (Day 1: Single oral dose Days 3 to 16: (14 Days) BID oral doses) or placebo for approximately 15 days. GSK2140944 dose in Cohort 3 will be decided on the safety data and available PK data from at least 12 subjects dosed at the Cohort 2
  Interventions: Drug: GSK2140944
- Cohort 3 - Placebo (Placebo Comparator): Subjects will be randomized in 12:4 ratio to receive either GSK2140944 bid or matching placebo for approximately 15 days
  Interventions: Drug: Placebo
- Cohort 4 - GSK2140944 2500 mg (Experimental): Subjects will be randomized in 12:4 ratio to receive either GSK2140944 (Day 1: Single oral dose Days 3 to 16: (14 Days) BID oral doses) or placebo for approximately 15 days. GSK2140944 dose in Cohort 4 will be decided on the safety data and available PK data from at least 12 subjects dosed at the Cohort 3
  Interventions: Drug: GSK2140944
- Cohort 4 - Placebo (Placebo Comparator): Subjects will be randomized in 12:4 ratio to receive either GSK2140944 bid or matching placebo for approximately 15 days
  Interventions: Drug: Placebo
- Cohort 5 - GSK2140944 TBD (Experimental): Subjects will be randomized in 6:2 ratio to receive either GSK2140944 (Day 1: Single oral dose Days 3 to 16: (14 Days) TID oral doses) or placebo for approximately 15 days. GSK2140944 dose in Cohort 5 will be decided on the safety data and available PK data from at least 12 subjects dosed at the Cohort 4
  Interventions: Drug: GSK2140944
- Cohort 5 - Placebo (Placebo Comparator): Subjects will be randomized in 6:2 ratio to receive either GSK2140944 TID or matching placebo for approximately 15 days
  Interventions: Drug: Placebo
- Cohort 6 - GSK2140944 TBD (Experimental): Subjects will be randomized in 6:2 ratio to receive either GSK2140944 (Day 1: Single oral dose Days 3 to 16: (14 Days) TID oral doses) or placebo for approximately 15 days. GSK2140944 dose in Cohort 5 will be decided on the safety data and available PK data from at least 6 subjects dosed at the Cohort 5
  Interventions: Drug: GSK2140944
- Cohort 6 - Placebo (Placebo Comparator): Subjects will be randomized in 6:2 ratio to receive either GSK2140944 TID or matching placebo for approximately 15 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK2140944 — GSK2140944 will be available as immediate release capsules of dose strength 100 mg and 500 mg
  Arms: Cohort 1 - GSK2140944 400 mg; Cohort 2 - GSK2140944 800 mg; Cohort 3 - GSK2140944 1500 mg; Cohort 4 - GSK2140944 2500 mg; Cohort 5 - GSK2140944 TBD; Cohort 6 - GSK2140944 TBD
Drug: Placebo — Matching placebo will be available
  Arms: Cohort 1 - Placebo; Cohort 2 - Placebo; Cohort 3 - Placebo; Cohort 4 - Placebo; Cohort 5 - Placebo; Cohort 6 - Placebo

SUMMARY:
This will be a randomized, placebo-controlled, single blind study to investigate the safety, tolerability and pharmacokinetic (PK) profile of GSK2140944 following repeat oral doses in healthy adult subjects. The study will include a Screening period (40 days), Treatment period (16 days) and a Follow-up period (26 to 30 days). A single dose will be administered on Day 1 for characterization of single dose PK, followed by twice-daily (BID) or thrice-daily (TID) dosing on Days 3 to 16. Subjects may only be randomized to one cohort per the randomization schedule. Up to 6 cohorts will be enrolled using a sequential panel. Subjects in Cohort 1 will receive GSK2140944 (6) and placebo (2). Subsequent cohorts will enroll 16 subjects such that 12 subjects will receive GSK2140944 and 4 subjects will receive placebo, per dose level according to the randomization schedule. Dose escalations are planned to run in successive weeks. Cohort 2 may begin dosing once subjects in Cohort 1 have completed 7 days of BID dosing, PK data is reviewed and safety data from at least 6 subjects is available. Each subsequent dose escalation will commence only when GSK2140944 safety data and available PK data of at least 12 subjects dosed at the previous dose level have been reviewed. The number of cohorts may be reduced or expanded if needed. The first planned dose is 400 milligram (mg) BID but may be modified based upon emergent PK, safety and tolerability data from ongoing clinical study BTZ115198 evaluating single and repeat intravenous (IV) doses of GSK2140944. The projected dose for Cohort 2 is 800 mg BID, Cohort 3 is 1500 mg BID, Cohort 4 is 2300 mg BID or 1500 mg TID and Cohort 5 and cohort 6 will be decided later. The planned maximum dose is 2500 mg TID but may be modified based upon emergent safety, tolerability and PK data. Doses of GSK2140944 or placebo will be administered following a moderate fat meal.

ELIGIBILITY:
Inclusion Criteria:

* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <=1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. - A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GlaxSmithKline (GSK) Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 60 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea. To confirm post-menopausal status, a blood sample for simultaneous follicle stimulating hormone (FSH) >40 MlU/ml and estradiol <40 pg/ml (<147 pmol/L) is confirmatory. Male subjects with female partners of child-bearing potential must agree to use the contraception methods. This criterion must be followed from the time of the first dose of study medication until the final follow-up visit.
* Body weight >=50 kg and body mass index (BMI) within the range 19 to 31 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening or positive Human Immunodeficiency Virus (HIV) antibody.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities.
* Any clinically significant central nervous system (e.g., seizures), cardiac, pulmonary, metabolic, renal, hepatic or gastrointestinal conditions or history of such conditions that, in the opinion of the investigator may place the subject at an unacceptable risk as a participant in this trial or may interfere with the absorption, distribution, metabolism or excretion of drugs.
* A screening or Day -2 urinalysis positive for protein or glucose (greater than "trace" findings of protein or glucose).
* A serum creatinine value between screening and Day -2 visit that is increased by more than 0.2 mg/dL (or 15.25 umol/L) changes.
* History of photosensitivity to quinolones and tendon rupture.
* Unwillingness to commit to avoid excessive exposure to sunlight which would cause a sunburn reaction from first dose up to and including the follow-up visit.
* A positive urine test for drugs of abuse or alcohol (or alcohol breath test) at screening or Day -2.
* History of drug abuse within 6 months of the study
* History of smoking or use of nicotine containing products within 3 months of screening, or a positive urine cotinine indicative of smoking at screening.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, or use of St. John's Wort within 14 days prior to the first dose of study medication. By exception, the volunteer may take paracetamol or acetaminophen (<=2 grams/day) up to 48 hours prior to the first dose of study medication. However, the Investigator and GSK study team can review medication on a case by case basis to determine if its use would compromise subject safety or interfere with the study procedures or data interpretation.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* History of sensitivity to heparin or heparin-induced thrombocytopenia (if the clinical research unit uses heparin to maintain intravenous cannula patency).
* Donation of blood in excess of 500 ml within 12 weeks prior to dosing.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice, pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices containing such products from 7 days prior to the first dose of study medication.
* Screening ECG: Heart rate <40 and >100 bpm for males and <50 and >100 bpm for females. PR Interval <120 and >220 msec, QRS duration <70 and >100 msec, QTcB or QTcF interval >450msec. Evidence of previous myocardial infarction (does not include ST segment changes associated with repolarization); any conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular (AV) block [2nd degree or higher], Wolf Parkinson White [WPW] syndrome), sinus pauses >3 seconds, non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats) or any significant arrhythmia which, in the opinion of the principal investigator and GSK medical monitor, will interfere with the safety of the individual subject.
* Screening holter monitoring shows one or more of the following: any symptomatic arrhythmia (except isolated extra systoles); sustained cardiac arrhythmias (such as atrial fibrillation or flutter, supraventricular tachycardia (SVT) [>10 consecutive beats]); sinus tachycardia (or SVT) >150 bpm; non-sustained or sustained ventricular tachycardia (defined as >=3 consecutive ventricular ectopic beats); any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher in an awake subject], WPW syndrome, other pre-excitation syndromes); symptomatic sinus pause or sinus pause >3 seconds - unless patient is straining, vomiting, or having some other type of hypervagal response; 300 or more supraventricular ectopic beats in 24 hours; 250 or more ventricular ectopic beats in 24 hours; Ischemia, diagnosed by a sequence of EKG changes that include flat or down sloping ST-segment depression >0.1 mV, with a gradual onset and offset that lasts for a minimum period of 1 minute. Each episode of ischemia must be separated by a minimum duration of at least 1 minute, during which the ST segment returns back to baseline (1x1x1 rule).
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* Neutrophil count <2000 cells per microliter (a single repeat is allowed for eligibility determination).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2012-10-17 (Actual); Primary Completion 2013-12-13 (Actual); Study Completion 2013-12-13 (Actual)

PRIMARY OUTCOMES:
GSK2140944 clinical safety data assessed as change from baseline in 12-lead ECG | Day 1, Day 4, Day 7, Day 10, Day 13, Day 16, Day 18 and at the Follow-up visit
  12-lead ECGs will be obtained at each timepoint using an ECG machine, after the subject has rested in a semi-supine position for at least 10 minutes
GSK2140944 clinical safety data from dual-lead cardiac monitoring | Day 1
  Continuous dual-lead cardiac monitoring will be obtained at each timepoints using an ECG machine
GSK2140944 clinical safety data assessed as change from baseline in clinical laboratory tests | Day -2 and pre-morning dose on Day 2, Day 5, Day 8, Day 11, and Day 14; on the morning of Day 17 and at the Follow-up visit
  Clinical laboratory assessments will include hematology, clinical chemistry, routine urinalysis and additional parameters
GSK2140944 clinical safety data assessed as by number of adverse events (AE) | Up to the Follow-up visit
  Safety and tolerability parameters will include recording of AEs, throughout the study
GSK2140944 clinical safety data assessed as change from baseline in blood pressure | Day -1, Day 1, Day 4, Day 7, Day 10, Day 13, Day 16, Day 18 and the Follow-up visit
  Vital sign measurements will be done in semi-supine position and will include systolic and diastolic blood pressure
GSK2140944 clinical safety data assessed as change from baseline in heart rate | Day -1, Day 1, Day 4, Day 7, Day 10, Day 13, Day 16, Day 18 and the Follow-up visit
  Vital sign measurements will be done in semi-supine position and will include pulse rate
Pharmacokinetic parameter: AUC(0-12) following single dose of GSK2140944 | Day 1
  Pharmacokinetic data will include area under the curve from time zero (pre-dose) to 12 hour post-dose (AUC(0-12)) following single dose of GSK2140944
Pharmacokinetic parameter: AUC(0-24) following single dose of GSK2140944 | Up to Day 2
  Pharmacokinetic data will include area under the curve from time zero (pre-dose) to 24 hour post-dose (AUC(0-24)) following single dose of GSK2140944
Pharmacokinetic parameter: AUC(0-t) following single dose of GSK2140944 | Up to Day 3
  Pharmacokinetic data will include area under the concentration-time curve from time zero (pre-dose) to last time of quantifiable concentration (AUC(0-t)) following single dose of GSK2140944
Pharmacokinetic parameter: AUC(0-infinity) following single dose of GSK2140944 | Up to Day 3
  Pharmacokinetic data will include area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC(0-infinity)) following single dose of GSK2140944
Pharmacokinetic parameter: Cmax following single dose of GSK2140944 | Up to Day 3
  Pharmacokinetic data will include maximum observed concentration (Cmax) following single dose of GSK2140944
Pharmacokinetic parameter: tmax following single dose of GSK2140944 | Up to Day 3
  Pharmacokinetic data will include time of occurrence of Cmax (tmax) following single dose of GSK2140944
Pharmacokinetic parameter: t1/2 following single dose of GSK2140944 | Up to Day 3
  Pharmacokinetic data will include terminal phase half-life (t1/2) following single dose of GSK2140944
Pharmacokinetic parameter: AUC(0-tau) following repeat dose of GSK2140944 | Day 14, Day 15 and Day 16
  Pharmacokinetic data will include area under the concentration-time curve over the dosing interval (AUC(0-tau)) following repeat dose of GSK2140944
Pharmacokinetic parameter: Cmax following repeat dose of GSK2140944 | Day 14, Day 15 and Day 16
  Pharmacokinetic data will include Cmax following repeat dose of GSK2140944
Pharmacokinetic parameter: tmax following repeat dose of GSK2140944 | Day 14, Day 15 and Day 16
  Pharmacokinetic data will include tmax following repeat dose of GSK2140944
Pharmacokinetic parameter: Ctau following repeat dose of GSK2140944 | Day 14, Day 15 and Day 16
  Pharmacokinetic data will include pre-dose (trough) concentration at the end of the dosing interval (Ctau) following repeat dose of GSK2140944
Pharmacokinetic parameter: Ro following repeat dose of GSK2140944 | Day 14, Day 15 and Day 16
  Pharmacokinetic data will include accumulation ratio (Ro) following repeat dose of GSK2140944
Pharmacokinetic parameter: AUC(0-8) following single dose of GSK2140944 | Day 1
  Pharmacokinetic data will include area under the curve from time zero (pre-dose) to 8 hour post-dose (AUC[0-8]) following single dose of GSK2140944

SECONDARY OUTCOMES:
To assess preliminary dose proportionality using PK parameter AUC(0-infinity) following single dose of GSK2140944 | Up to Day 3
  Preliminary dose proportionality will be assessed using PK parameter (AUC(0-infinity)) following single dose of GSK2140944
To assess preliminary dose proportionality using PK parameter Cmax following single dose of GSK2140944 | Up to Day 3
  Preliminary dose proportionality will be assessed using PK parameter Cmax following single dose of GSK2140944
To assess preliminary dose proportionality using PK parameter AUC(0-tau) following repeat doses of GSK2140944 | Day 14, Day 15 and Day 16
  Preliminary dose proportionality will be assessed using PK parameter (AUC(0-tau) following repeat doses of GSK2140944
To assess preliminary dose proportionality using PK parameter Cmax following repeat doses of GSK2140944 | Day 14, Day 15 and Day 16
  Preliminary dose proportionality will be assessed using PK parameter Cmax following repeat doses of GSK2140944
To examine extent of accumulation using PK parameter Ro using AUC(0-tau) following repeat doses of GSK2140944 | Day 14, Day 15 and Day 16
  Accumulation ratio will be assessed using PK parameter AUC(0-tau) following repeat doses of GSK2140944
To examine extent of accumulation using PK parameter AUC(0-tau) following single dose of GSK2140944 | Day 1
  Accumulation ratio will be assessed using PK parameter AUC(0-tau) following single dose of GSK2140944
To examine the extent of time invariance using repeat dose AUC(0-tau) | Day 14, Day 15 and Day 16
  The extent of time invariance will be assessed using PK parameter AUC(0-tau) following repeat dose
To examine the extent of time invariance using single dose AUC(0-infinity) | Up to Day 3
  The extent of time invariance will be assessed using PK parameter AUC(0-infinity) following single dose
To assess achievement of steady-state following repeat oral doses of GSK2140944 | Day 14, Day 15 and Day 16
  Achievement of steady-state will be assessed using trough concentrations at the end of the dosing interval (Ctau) collected at pre-morning dose on Days 14 and 15 (together with pre-morning dose Ctau on Days 16 from the full PK profiles on Day 16).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Tiffany C, Dumont EF, Hossain M, Srinivasan M, Swift B. Pharmacokinetics, safety, and tolerability of gepotidacin administered as single or repeat ascending doses, in healthy adults and elderly subjects. Clin Transl Sci. 2022 Sep;15(9):2251-2264. doi: 10.1111/cts.13359. Epub 2022 Jul 13. PMID 35769034
- See also: Results for study 116778 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/116778?search=study&search_terms=116778#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 116778 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116778 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116778 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116778 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116778 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116778 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116778 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register